CLINICAL TRIAL: NCT00818402
Title: Treatment of Non-small Cell Lung Cancer -Effects on Quality of Life and Symptom Control
Brief Title: Non-small Cell Lung Cancer and Quality of Life
Acronym: SILKE
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Maria Silvoniemi, MD, University of Turku
Other Study IDs: SILKE-ETMK:47/180/2008
Record Dates: First submitted 2009-01-05; First posted 2009-01-07 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Quality of life; symptoms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-small cell lung cancer patients

SUMMARY:
The principal objective is to study clinical observations, symptoms and quality of life of non-small-cell lung cancer (NSCLC) patients undergoing specific non-operative treatment for cancer, including chemotherapy and radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with verified NSCLC
* after the NSCLC diagnosis has been confirmed prior to first chemotherapy or radiotherapy
* Finnish speaking patients
* aged 18 years or more
* Written informed consent has to be signed

Exclusion Criteria:

* Patients not consenting to participate in the study
* patients not able to communicate sufficiently
* cancer type is other than non-small-cell lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients treated in the clinic of respiratory medicine in Turku, Finland
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2008-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)